CLINICAL TRIAL: NCT07090252
Title: Clinical and Radiographic Evaluation of Zinc Oxide-eugenol and Zinc Oxide With Neem as Obturating Materials in Primary Mandibular Molars Pulpectomy for 5-7 Year-Old Children: A Randomized Clinical Trail
Brief Title: Comparison of ZOE vs ZON in Primary Mandibular Molars Pulpectomy of 5-7-Year-Olds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tasneem Ali Osman Ali, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRP-ZOE Vs ZON
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I zinc oxide with Neem (Experimental): Neem and zinc oxide powder have been improved as a theraputic agents with high antibacterial, antioxidant, and enzyme-inhibiting properties against microorganisms resistant to antibiotics.Neem contains many chemically diverse and structurally complex phytochemicals, such as limonoids, flavonoids, phenols, catechins, gallic acid,polyphenols, and nimbins which contribute to their different pharmacological activities.
  Interventions: Other: Group I zinc oxide Neem
- Group II zinc oxide -eugenol (Experimental): zinc oxide eugenol is a mixture of zinc oxide (powder) and eugenol (liquid). Zinc oxide and eugenol (ZOE) paste is a standard in dentistry among the pastes used in the pulp therapy of primary teeth.
  Interventions: Other: Group II zinc oxide eugenol

INTERVENTIONS:
Other: Group I zinc oxide Neem — preperation: 1\ A standardized access cavity procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, a sharp spoon excavator will remove coronal pulpal tissues then will remove radicular pulp by barbed broach then will be used K files for chemo mechanical preparation (size 15,20,25) with saline (2%) irrigation to remove necrotic pulp tissues then all the canals will be dried using paper points. 2\ After complete excavation of all pulp tissue, saline irrigation is done then the canals will be obturated zinc-oxide with Neem ( Zinc oxide powder(Prime Dental Pvt. Ltd.Thane, Maharashtra, India) and 100% Neem oil with mixing ratio of 1:3 will be mixed on a glass slab with a stainless- steel spatula) and then the rest of the pulp chamber will be filled with Zinconol. (reinforced zinc oxide eugenol)3\ Tooth will be restored with stainless steel crown.
  Arms: Group I zinc oxide with Neem
Other: Group II zinc oxide eugenol — preperation: 1\ A standardized access cavity procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, a sharp spoon excavator will remove coronal pulpal tissues then will remove radicular pulp by barbed broach then will be used K files for chemo mechanical preparation (size 15,20,25) with saline (2%) irrigation to remove necrotic pulp tissues then all the canals will be dried using paper points 2\ After complete removed of coronal and radicular pulp zinc oxide eugenol will be manipulated in the ratio of 3:1 (powder: liquid) to obtain semisolid mix.This mix will be placed in the canals. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by the application of Zinconol.3\ Tooth will be restored with stainless steel crown.
  Arms: Group II zinc oxide -eugenol

SUMMARY:
The goal of this clinical trial is to evaluation of Zinc oxide-eugenol compared to Zinc oxide with Neem as obturating materials in primary mandibular molars pulpectomy for 5-7 Year-Old Children.The main question(s)it aim to answer : Could the clinical and radiographic success of a mixture of zinc oxide with Neem oil be comparable with Zinc oxide-eugenol paste in pulpectomy of primary mandibular molars?

DETAILED DESCRIPTION:
Dental caries is a global public health issue that mostly affects children in their early childhood, negatively impacting both their oral and overall health .The primary teeth with pulpal and periapical problems, should be kept until their natural exfoliation because their early loss could result in undesired abnormalities in the dentition later on . The complex root canal morphology, intrinsic physiologic root resorption, close proximity to the permanent successors, difficulty obtaining good radiographic views of the tooth apices, complex diagnosis due to the patient's immaturity, requirement for behavioral guidance of pediatric patients, technique selection, and root filling material selection make pulpectomy in primary teeth still controversial .When the pulp becomes irreversibly infected or necrotic, root canal therapy is recommended for children. The most common root canal filling material for primary teeth is zinc oxide eugenol (ZOE). However, it has some drawbacks, including slow resorption, periapical tissue irritation, and bone and cementum necrosis, which can result in anterior cross bite, palatal eruption, or ectopic eruption of a succedaneous tooth. As a result, ongoing research is required to find the ideal obturation material.To ensure the success of the endodontic treatment, various materials with good antimicrobial properties are used as root canal filling materials in primary teeth Phytodentistry has become a growing field in dentistry. It refers to the use of medicinal plants and their products to treat disease, either directly or indirectly. ZOE has been attempted with a variety of chemicals to improve its characteristics and success rate, however neither the success rate nor the material's resorbability were improved when compared to ZOE alone.Eugenol irritates the periapical area and solidifies into hard mass when combined with ZnO powder. Neem belongs to the family Meliaceae, also known as Azadirachta indica, is a plant that originated in India and now thrives in tropical and subtropical regions worldwide. It is highly valued for its therapeutic benefits. Neem contains a variety of biologically active compounds, including alkaloids, flavonoids, triterpenoids, phenolic compounds, carotenoids, steroids, and ketones. It has strong antimicrobial properties that can help manage and prevent various infections.This can aid in pharmacovigilance by monitoring and managing antibiotic and antimicrobial side effects. It has many medical uses such as immunoregulatory, antifungal, antihyperglycemic, antiulcer, antimalarial, anti inflammatory, antibacterial, antiviral, and antioxidant

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5-7 years with infected primary molars.
2. Deep carious lesion.
3. History of spontaneous pain
4. Parent written informed consent.

Exclusion Criteria:

1. Medically compromised children
2. Children with a history of allergic reaction to the components of the tested material
3. Children who had non restorable teeth
4. Teeth with less than two third of root length
5. Extensive internal or external root resorption
6. Unable to attend follow-up visits

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | [Time Frame: follow-up: T(Time):12months interval T0:0 T1:3month T2:6month T3:9month T4:12month]
  1. Absence of pain method of measurement: verbal question to patient/parent Outcome measuring unit: Binary(Yes/No)
  2. Absence of tenderness to percussion method of measurement: percussion test by the back of the dental mirror Outcome measuring unit: Binary(Yes/No)
  3. Absence of swelling and sinus tract method of measurement: Visual and Clinical examination Outcome measuring unit: Binary(Yes/No)
  4. Absence of mobility:
  method of measurement: Mobility test by using two single-ended instruments(dental mirror and probe) Outcome measuring unit: Binary(Yes/No)

SECONDARY OUTCOMES:
Radiographic Success | [Time Frame: follow-up: T(Time):12months interval T0:0 T2:6month T4:12month]
  1. Absence or reduction in the size of periapical radiolucency Method of measurement: Visual interpretation for intra-oral periapical radiograph Outcome measuring unit: Binary(Yes/No)
  2. Absence or reduction in the size of furcation radiolucency Method of measurement: Visual interpretation for Intra-oral periapical radiograph Outcome measuring unit: Binary(Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Adel Elbardissy, Prof Doctor, Study Director — Cairo University
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, El-manial, Egypt

IPD SHARING:
Plan to Share IPD: No